CLINICAL TRIAL: NCT04362280
Title: Teens Committed to Health Through Activity, Relationships, and Good Eating (Take CHARGE!)
Brief Title: Teens Committed to Health Through Activity, Relationships, and Good Eating
Acronym: Take CHARGE!
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Craig A Johnston, Associate Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001135
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ReCHARGE (Experimental): intervention intensity is increased through: the creation of family groups, greater involvement of school staff, separate lessons for females, health screeners will be home and families are invited to a nutrition counseling session with a registered dietitian.
  Interventions: Behavioral: ReCHARGE
- Treatment as Usual (TAU) (Active Comparator): PE class as usual which consisted of choice time.
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: ReCHARGE — During their PE class, all participants (both arms) participate in an intensive lifestyle intervention with established efficacy among this population for the academic fall semester. The following semester, participants are randomized to different treatment arms. ReCHARGE increases the intensity of treatment provided in the first semester by increasing social support and addressing common barriers youth have to adhering to intervention.
  Arms: ReCHARGE
Behavioral: TAU — PE class as usual led by PE teacher.
  Arms: Treatment as Usual (TAU)

SUMMARY:
This study will evaluate the preliminary efficacy of a school-based weight management program for underserved adolescents. The program was designed with a phased treatment structure to provide more intensive treatment to participants who do not respond to treatment initially. Specifically, this study aims to examine differences in zBMI over time between students who do not respond to the first semester and receive more intensive treatment in the second semester, responders to first semester who receive more intensive treatment in the second semester, non-responders to the first semester who receive usual treatment in the second semester, and responders who receive usual treatment in the second semester at the end of the second semester, 1 year follow-up, and 2 year follow-up.

DETAILED DESCRIPTION:
Childhood obesity has reached epidemic proportions. Schools have been identified as a focal point for intervention because children spend almost half their day in school. On average, school-based interventions have shown modest short-term improvements in weight outcomes. However, considerable individual variation is found within treatments. Current clinical guidelines for childhood obesity recommend a staged treatment approach in which every few months treatment plans are reevaluated based on an individual's progress toward weight outcomes. When an individual doesn't sufficiently progress toward outcome goals, his/her treatment is escalated to be more individualized, include more structure, and greater social support. This method parallels a treatment paradigm used in other areas of medical treatment in which medication type and dose are altered when an individual does not respond to initial care. Obesity treatment provided in the school setting does not follow a similar structure of care. Despite the recognized variation between individuals, school-based obesity interventions are typically evaluated by mean changes in weight outcomes over time. Although this is sufficient to evaluate the efficacy of a program, it does not identify individuals who are not responsive to treatment. Following clinical best practices, it is likely that treatment needs to be escalated for those who do not respond to initial treatment. Currently no escalated treatment options, like that provided in clinical settings, are available in schools. This is a critical gap given the immense individual variability to treatment response and pediatric tracking of BMI. This study will develop and evaluate an escalated school-based treatment for individuals resistant to initial treatment, called Take CHARGE! (Teens Committed to Health through Activity, Relationships, and Good Eating). Specifically, a pilot randomized control trial will A.) examine differences in zBMI between Take CHARGE and a treatment as usual condition over an academic school semester among low SES, racial/ethnic minority youth resistant to initial treatment, and will B.) determine the proportion of students resistant to school-based behavioral obesity treatment. Understanding the proportion of children who are resistant to school-based intervention is a critical first step in treating this high-risk group of children.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10-17 years old
* Student enrolled in a Physical Education (PE) class at the YES Prep Brays Oak Campus during either the 2018-2019 or 2019-2020 school year
* provides written parental consent and student assent

Exclusion Criteria:

* Is pregnant or becomes pregnant during the study.
* Is unable to participate in PE class for more than 5 consecutive school days.
* Does not meet all of the inclusion criteria listed above

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 392 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Standardized BMI | up to 2 years
  Examine zBMI over the course of the intervention between study arms

SECONDARY OUTCOMES:
Social Network | up to 6 months
  students asked to list their friends in the class

OTHER OUTCOMES:
Carotenoid levels | up to two years
  Veggie Meter carotenoid measures

CONTACTS AND LOCATIONS:
Overall Officials: Craig A Johnston, PhD, Principal Investigator — University of Houston
Locations (1):
- YES Prep Brays Oaks, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arlinghaus KR, O'Connor DP, Ledoux TA, Hughes SO, Johnston CA. A staged approach to address youth unresponsive to initial obesity intervention: a randomized clinical trial. Int J Obes (Lond). 2021 Dec;45(12):2585-2590. doi: 10.1038/s41366-021-00940-0. Epub 2021 Aug 20. PMID 34417553